CLINICAL TRIAL: NCT06975059
Title: Using the NUSHU Shoe to Analyze Gait Balance and Vibrotactile Feedback in Early, Moderate and Advanced PD Patients and Healthy Controls
Brief Title: Novel Shoe Device NUSHU to Measure Gait Analysis in Parkinson's Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-05027451
Record Dates: First submitted 2025-05-08; First posted 2025-05-16 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Parkinson's Disease (PD)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Parkinson's Disease (Early) (Experimental): The early PD group will be those within 3 years of diagnosis. Each group will be administered the same administration of 4 visits, with 3 of the visits wearing the shoes with and without vibration in clinic.
  Interventions: Device: NUSHU shoe
- Parkinson's Disease (Moderate) (Experimental): The moderate PD group will be those with 4-7 years of diagnosis. Each group will be administered the same administration of 4 visits, with 3 of the visits wearing the shoes with and without vibration in clinic.
  Interventions: Device: NUSHU shoe
- Parkinson's Disease (Advanced) (Experimental): The advanced PD group will be those with at least 8 years of diagnosis. Each group will be administered the same administration of 4 visits, with 3 of the visits wearing the shoes with and without vibration in clinic.
  Interventions: Device: NUSHU shoe
- Healthy Controls (Active Comparator): Healthy controls will include those without any neurological disease or other significant gait impairment. Each group will be administered the same administration of 4 visits, with 3 of the visits wearing the shoes with and without vibration in clinic.
  Interventions: Device: NUSHU shoe

INTERVENTIONS:
Device: NUSHU shoe — The NUSHU shoe, created by Magnes AG, can measure real-time detection of gait analysis while providing vibrotactile stimulus to the study participant through machine learning sensors. This may provide a feedback mechanism that acts as therapy for gait difficulties.

SUMMARY:
Gait changes in Parkinson's disease are complex, variable, and difficult to detect during short clinic assessments. The aim of this study is to collect gait measurements in Parkinson's patients through sensors in a novel shoe device, NUSHU by Magnes AG. The shoe additionally provides vibrational feedback that can potentially help gait difficulties experienced by Parkinson's patients.

ELIGIBILITY:
Parkinson's Disease:

Inclusion Criteria:

1. Male or female ≥ 18 years of age.
2. A diagnosis of Parkinson's disease
3. Able to give written informed consent (as determined by the investigator)
4. Can converse in English and read and perform all study activities
5. Has willingness and ability to comply with study requirements

Exclusion Criteria:

1. Diagnosis of an atypical parkinsonism syndrome, drug-induced parkinsonism, essential tremor, or other diagnoses that explain movement symptoms other than PD
2. A diagnosis of significant CNS disease other than PD such as stroke, multiple sclerosis, epilepsy
3. Persons with disorders other than PD significantly affecting gait as determined by the investigator
4. History of MRI brain scan indicative of clinically significant abnormality as determined by the investigator
5. Inability to wear interventional device
6. Unable to ambulate independently at least with assistive walking device but without additional person assistance
7. Pregnant or planning pregnancy within study timeframe
8. Montreal Cognitive Assessment (MoCA) score < 22 at screening
9. Resides in a nursing home or assisted care facility

Healthy Controls:

Inclusion Criteria:

1. Male or female ≥ 18 years of age.
2. No neurological disease or other significant gait impairment as deemed by the study investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Mean Score of Comfort Level of Device in Satisfaction Survey | At Safety Follow Up (Week 18)
  The satisfaction survey contains 2 demographic questions and 5 questions about participant satisfaction completed at end of study participation. The comfort level of the device question is the following: How would you rate the comfort level of the device? The scale is 0, 1, 2, 3, 4, 5, with 0 meaning most uncomfortable and 5 meaning most comfortable. Mean score for each individual question will be provided.
Mean Score of Ease of Using Device in Satisfaction Survey | At Safety Follow Up (Week 18)
  The satisfaction survey contains 2 demographic questions and 5 questions about participant satisfaction completed at end of study participation. The comfort level of the device question is the following: How easy was it to use the device? The scale is 0, 1, 2, 3, 4, 5, with 0 meaning very easy and 5 meaning very difficult. Mean score for each individual question will be provided.
Ratio of Participants Who Completed Study to Total Number of Participants Enrolled | Through study completion, 18 weeks
  We would like to measure the retention rate to assess feasibility. The lowest ratio would be 0, and the highest ratio would be 1.

SECONDARY OUTCOMES:
Mean Change from Baseline to Week 12 in TUG test | At Baseline and In 12 Weeks
  Timed Up and Go test assesses mobility, balance, walking ability, and fall risk in older adults by measuring how quickly the patient can stand up, walk 10 feet, turn around, walk back, and sit down. The score is the amount of time taken in seconds. There is no highest nor lowest score. The higher the time, the more problems the patient has with gait and requires gait aid.
Mean Change from Baseline to Week 12 in FOG Questionnaire | At Baseline and In 12 Weeks
  Freezing of Gait questionnaire assesses FOG severity unrelated to falls, FOG frequency, gait disturbances, and relationship to clinical features associated with gait and motor aspects in Parkinson's patients. The score ranges from 0 to 24, and high scores correspond to more severe FOG.
Mean Change from Baseline to Week 12 in MDS-UPDRS III | At Baseline and In 12 Weeks
  The Movement Disorder Society (MDS)-Unified Parkinson's Disease Rating Scale (UPDRS) Part III (motor examination; to be completed in the on-medication state) has instructions for the rater to give or demonstrate to the participant; it is completed by the investigator. Each question has a 0-4 rating scale. The total scores range from 0 to 132, with higher scores indicate increased severity.
Mean Change from Baseline to Week 12 in Stride Time | At Baseline and In 12 Weeks
  The NUSHU shoe measures the stride time: the time elapsed between the first contact of two consecutive footsteps of the same foot. This time is collected in seconds.
Mean Change from Baseline to Week 12 in Stride Length | At Baseline and In 12 Weeks
  The NUSHU shoe measures the stride length: the distance covered between the same spot where one foot hits the ground and the next time the same foot hits the ground again. This distance is collected in meters.
Mean Change from Baseline to Week 12 in Swing Time | At Baseline and In 12 Weeks
  The NUSHU shoes measure the swing time: the amount of time the foot spends off the ground in the gait cycle, defined by the time from toe off to heel strike of the same foot. The time is collected in seconds.
Mean Change from Baseline to Week 12 in Stance Time | At Baseline and In 12 Weeks
  The NUSHU shoes measure the stance time: the duration of the time between heel strike and toe off of the same foot. This time is collected in seconds.
Mean Change from Baseline to Week 12 in Velocity | At Baseline and In 12 Weeks
  The NUSHU shoes measure the velocity: mean in-plane velocity of each gait cycle (m/s).
Mean Change from Baseline to Week 12 in Cadence | At Baseline and In 12 Weeks
  The NUSHU shoes measure the cadence: number of strides per minute.
Mean Change from Baseline to Week 12 in Swing Phase | At Baseline and In 12 Weeks
  The NUSHU Shoes measure the swing phase: ratio of swing time with respect to gait cycle duration.
Mean Change from Baseline to Week 12 in Stance Phase | At Baseline and In 12 Weeks
  The NUSHU shoes measure the stance phase: ratio of stance time with respect to gait cycle duration.

CONTACTS AND LOCATIONS:
Overall Officials: Harini Sarva, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No